CLINICAL TRIAL: NCT00735111
Title: Do Self-Rated Karnofsky Performance Status (KPS) Scores Correlate With Health-Care-Provider-Rated Scores?
Brief Title: Do Self-Rated Performance Status Scores Correlate With Health-Care-Provider-Scores?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: QOL-001
Record Dates: First submitted 2008-08-13; First posted 2008-08-14 (Estimated); Last update posted 2013-01-17 (Estimated); Status verified 2013-01

CONDITIONS: Cancer
Keywords: QOL; Quality of Life; KPS; Karnofsky Performance Status; Cancer
MeSH Terms: conditions — Neoplasms | interventions — Karnofsky Performance Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Karnofsky Performance Status Score (Experimental)
  Interventions: Other: Karnofsky Performance Status Score

INTERVENTIONS:
Other: Karnofsky Performance Status Score — Karnofsky Performance Status scores will be independently completed by both the patient and their health-care provider at each routine clinic visit.
  Other Names: Performance Status Scale

SUMMARY:
The purpose of this study is to determine if patients are able to self-rate their physical abilities and how these ratings compare to the ratings of their health-care provider.

DETAILED DESCRIPTION:
The Karnofsky Performance Scale (KPS) is a highly validated and essential measuring tool across the cancer population. The scale relates to purely physical ability and covers 11 stages, ranging from normal health to death, with each stage scored as a percentage. The score is determined by the health-care provider and is based on observation and narrative patient descriptions. The purpose of this study is to compare the scores rated by the health-care provider to the scores that patients assign to themselves.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of brain or spinal tumor.
* Receiving medical care under the supervision of the Principal Investigator.
* Written informed consent.

Exclusion Criteria:

None.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2008-02; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
To determine the correlation between self-rated and health-care-provider-rated Karnofsky Performance Status scores. | 2 Years

CONTACTS AND LOCATIONS:
Overall Officials: Erin M Dunbar, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States